CLINICAL TRIAL: NCT06424808
Title: Pilot Study for the Validity of a Content-based Information Provision Tool Aimed at Improving the Hospitalization Experience of Liver Transplant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Taerim Kim, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-04-078-001
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Liver Transplantation; Inpatients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): 1. The group assigned as the control group will receive information in the same manner as it is currently provided to patients.
  2. A survey related to patient experience evaluation will be conducted before discharge. The survey will take about 10 minutes.
  3. The control group will undergo two interviews, one during hospitalization and one before discharge. Each interview will last approximately 30 minutes. Interviews will be recorded or transcribed, and the recordings will be used until the research objectives are met, after which they will be disposed of.
- Experimental Group (Experimental): 1. The group assigned as the experimental group will receive information in the same manner as it is currently provided to patients, with the addition of a brochure provided once when moving to a general ward after surgery. The brochure can then be used freely.
  2. A survey related to patient experience evaluation will be conducted before discharge. For the experimental group, an additional survey regarding the provided brochure will be included. The survey will take about 15 minutes.
  3. The experimental group will undergo two interviews, one during hospitalization and one before discharge. Each interview will last approximately 30 minutes. Interviews will be recorded or transcribed, and the recordings will be used until the research objectives are met, after which they will be disposed of.
  Interventions: Other: Consolidating content on a single website and providing access to it via QR codes in a brochure format

INTERVENTIONS:
Other: Consolidating content on a single website and providing access to it via QR codes in a brochure format — The group assigned to the experimental group will receive information in the same manner as current patients do, with the addition of receiving a brochure once when moving to a general ward after surgery. Afterward, they are free to use the brochure. The control group will receive information only in the manner currently provided to patients.
  Arms: Experimental Group

SUMMARY:
The investigators aim to evaluate the improvement of the inpatient experience and the usability of a content-based tool (a brochure). This involves consolidating video content for inpatients on a single website and providing access to it via QR codes in a brochure format.

[Patients] Considering this as a pilot study, the investigators plan to recruit around 30 participants. Both the experimental and control groups will receive standard care and information, with the experimental group additionally receiving the brochure. Random assignment will be used for the experimental and control groups. Surveys and interviews will be conducted to assess changes in patient experience and usability before and after providing the brochure.

[Medical Staff] Among the medical staff involved in the liver transplant surgical process, researchers will select participants based on their degree of involvement with the intervention subjects. After obtaining their consent, interviews will be conducted concerning patient experiences and the brochure.

ELIGIBILITY:
Inclusion Criteria:

[Patients]

* Adults aged 18 and over
* Patients who are scheduled to undergo or have undergone liver transplant surgery
* Recruited through a call for research participants and have consented to participate in this study

[Medical Staff]

* Adults aged 18 and over
* Medical staff at Samsung Medical Center involved in the post-liver transplant treatment process

Exclusion Criteria:

[Patients]

* Individuals who have not consented to participate in this study
* Individuals whose health condition makes it difficult to participate in the intervention
* During the research period, the researcher will check if the brochure content has been shared during surveys or interviews with the research participants (information dissemination). If information dissemination is confirmed, the participant will be excluded from the study.

[Medical Staff]

* Individuals who have not consented to participate in this study
* Medical staff not involved in the liver transplant treatment process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-21 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Inpatient Experience 1 | During the intervention
  Inpatient Experience Evaluation Score, which ranges from a minimum of 0 to a maximum of 100 points, with higher scores indicating better patient experiences.
Inpatient Experience 2 | During the intervention
  Analysis of survey response trends and frequencies between the experimental and control groups
Inpatient Experience 3 | Patient: During the intervention and after intervention(Two times)/Medical staff: During the study period
  Qualitative research through interviews

SECONDARY OUTCOMES:
Informational value of the intervention tool | During the intervention
  Asking informational value of the intervention tool from survey and interview
Usability value of the intervention tool | During the intervention
  Survey uses 'System Usability Scail' which ranges a minimum of 0 to a maximum of 100 points, with higher scores indicating better usability. Also related question will be asked by intervew.
Regarding utilization of the intervention tool | During the intervention
  A survey and interview on the experience of utilization during hospitalization
Areas for improvement | During the intervention
  A survey and interview on the advice for improvement

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the start to the end of the study
Access Criteria: Shared with all researchers approved by the IRB